CLINICAL TRIAL: NCT02200809
Title: MR-guided Focal Laser Ablation of the Prostate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Canisius-Wilhelmina Hospital (Other); Ziekenhuisgroep Twente (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010/185
Record Dates: First submitted 2014-07-21; First posted 2014-07-25 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2018-04

CONDITIONS: Prostate Cancer; MRI; Focal Laser Ablation
Keywords: MR-guided therapy; Focal laser ablation; Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MR-guided focal laser ablation (Experimental)
  Interventions: Device: MR-guided focal laser ablation

INTERVENTIONS:
Device: MR-guided focal laser ablation

SUMMARY:
Purpose of the investigators study is to determine the short and medium term histological cancer control of focal therapy using MR-guided focal laser ablation therapy in the treatment of localised prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed and biopsy proven prostate cancer
* Intermediate risk patients (PSA <= 20 ng/mL, Gleason ≤ 7, T2b)
* No previous treatment for prostate cancer
* Cancer lesion located at least 1 cm away from the neurovascular bundle according to Multimodality MR images
* Signed informed consent by patient
* Age 18 years or older
* Signed screening form (to determine exclusion for metal device/foreign bodies/claustrophobia)

Exclusion Criteria:

* Impossibility to obtain a valid informed consent
* Patients unable to undergo MR imaging, including those with contra-indications
* Contra-indications to MR guided focal laser therapy (colitis ulcerosa, rectal pathology or abdomino perineal resection)
* Metallic hip implant or any other metallic implant or device that distorts local magnetic field and compromises the quality of MR imaging
* Patients with evidence for nodal or metastatic disease
* Patients with an estimated Glomerular Filtration Ratio (eGFR) < 40 mL/min/1.73 m2

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-07 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Disease free survival | 36 months.
  The short and medium term histological cancer control defined as the percentage of patients with disease free survival according to the pathological MR-guided biopsy results after 36 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jurgen Futterer, MD, PhD, Principal Investigator — Radboud University Nijmegen Medical Center
Locations (3):
- Netherlands (3):
  - Radboud University Medical Center, Nijmegen, Gelderland
  - Canisius Wilhelmina Hospital, Nijmegen, Gelderland
  - Ziekenhuisgroep Twente, Hengelo, Overijssel